CLINICAL TRIAL: NCT01113242
Title: Characteristics of Cognitive Decline During Parkinson's Disease in the Elderly
Brief Title: Neuropsychological Assessment of Cognitive Decline in Patients With a Definite Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 4682
Record Dates: First submitted 2010-04-27; First posted 2010-04-29 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2010-11

CONDITIONS: Parkinson Disease Dementia
Keywords: Parkinson Disease Dementia; Observational; Case control; Neuropsychological assessment
MeSH Terms: interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- A:: Patients with idiopathic PD and with MMSE < à 26
  Interventions: Other: Neuropsychological Assessment
- B:: Patients with idiopathic PD and with MMSE ≥ à 26
  Interventions: Other: Neuropsychological Assessment

INTERVENTIONS:
Other: Neuropsychological Assessment — Included patients had clinically idiopathic PD, were over 65 years old and presented with a cognitive complain. A detailed registration of clinical history (including review of motor, cognitive, and neuropsychiatric symptoms, comorbid medical conditions, and medications) and neurologic examination was performed. Exclusion criteria included other conditions than PD that could contribute substantially to the subject's motor and/or cognitive impairment, including neurologic and major psychiatric disorders ( delirium,…) affecting the cognitive functions. Patients with major cognitive impairment (i.e. Mental State Examination (MMSE) <16/30) were also excluded.). Neuropsychological assessment explores working memory, episodic memory ,verbal fluency, executive functions and visuo constructive functions.

SUMMARY:
Cognitive disorders in Parkinson's disease (PD) are not as obvious as cognitive disorders in Alzheimer disease and their diagnosis tends to be delayed. If neuropsychological assessment of cognitive decline in Parkinson's disease is well established, the thresholds of cognitive testing corresponding to a dementia are unknown. Recently, new diagnosis criteria of dementia associated with PD have been proposed by the movement disorder society. In this study two groups of patients with idiopathic PD will be separated and compared according to their Mini Mental State Examination (MMSE) score (upper or lower than 26). Included patients will have clinically idiopathic PD, will be over 65 years old and will present cognitive complain. Cognitive and mood disorders as well as motor symptoms will be assessed using validated scales and a neuropsychological assessment dispatched in two visits will be performed . Differences in the distribution of data from the two groups of patients will be assessed in statistically analysis with non parametric tests. The purpose of this study is to determine the most effective tests and their threshold value corresponding to a pathological cognitive decline.

ELIGIBILITY:
Inclusion Criteria:

* MMSE ≥ 16
* impact of cognitive disorders in daily living
* criteria of the UKPDSBB for PD
* steady state in PD
* benign delusions or treated psychosis are tolerated
* informed consent obtained

Exclusion Criteria:

* dementia from other origin than PD
* cognitive decline without impact on daily living
* MMSE < 16
* delirium in the last 3 months
* Severe Depression
* Central Anticholinergic medication
* inability to perform the cognitive testing
* major cerebrovascular disease
* inability to give an informed consent (patients with protective measures)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients with idiopathic PD are issued from an ambulatory following at the department of Geriatrics
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2010-06 (Actual); Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michèle Kiesmann, MD, Principal Investigator — University Hospital, Strasbourg, France
Locations (1):
- Service de Gériatrie, Hôpital de la Robertsau, Hôpitaux Universitaires de Strasbourg, Strasbourg, France